CLINICAL TRIAL: NCT03373851
Title: Usability and Satisfaction Evaluation of Sufentanil Sublingual Patient-Controlled Analgesia After Elective Surgery With Moderate-to-Severe Postoperative Pain
Brief Title: Sublingual Sufentanil PCA Usability for Postoperative Pain (Zalviso® System)
Acronym: USE-SSPC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0511
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Trauma; Surgery
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Zalviso: Patient willing to participate to the study, and scheduled for major functional surgery (arthroplasty, valgisation osteotomy, DIEP flap surgery, total body lift procedures) will be consented to use the Zalviso device in postoperative period as a main analgesia method.
  Interventions: Device: Zalviso Device

INTERVENTIONS:
Device: Zalviso Device — The Zalviso device will be provided immediately before the Post anesthesia care unit (PACU) discharge. Patients will be queried every day during three postoperative days for the ability to use the device, their satisfaction, the level of pain, and the incidence of side effects. There will be no changes in usual care.
  In the end of this study ward nurses carrying Zalviso patients will be asked to provide their usability and satisfaction evaluation for Zalviso device management. Physical therapist will be asked to provide their satisfaction regarding patients' ability to follow physical therapy program.

SUMMARY:
Intravenous patient-controlled analgesia (iv-PCA) is the gold standard for the treatment of moderate to severe postoperative pain. It is used in more than 20% of cases after major surgery. Well known disadvantages of this method include the need of intravenous line (invasive, infection risk), the risk of pump programming error, possible delay for ambulation/barrier for enhanced rehabilitation programmes, and time/resource demanding (the need of preparation and installation). Sublingual sufentanil based PCA (Zalviso®) addresses cited issues. The safety and analgesia efficiency of this system is well described. However, the usability and satisfaction of Zalviso® varies depending on clinical settings. The goal of this study is to evaluate the usability and satisfaction of patients, nurses, and physical therapists using Zalviso® System during the first 72 hours in the settings of Enhanced Recovery After Surgery protocol after major interventions associated with moderate to severe postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* 16 <BMI <40
* ASA I and II
* Patient with traumatic functional surgery - Knee and hip arthroplasty, shoulder surgery, tibial osteotomy / femoral osteotomy; or plastic and aesthetic surgery with volume correction of more than 30% of body surface area (bodylift), DIEP, DLA.
* Patient who should theoretically benefit of a postop self-controlled analgesia of morphine for 72 hours on average
* Patient informed of the modalities of the study with delivery of an information leaflet
* Free and informed consent collection

Exclusion Criteria:

* Patient refusing to participate in the study
* Language barrier
* Hypersensitivity to sufentanil,
* Respiratory failure
* Renal insufficiency (GFR <30 ml / min)
* Epilepsy not controlled by treatment
* Psychic and mental illness not controlled by treatment
* Hepatocellular insufficiency (TP <50%)
* Heart failure (LVEF <50%)
* patients with chronic pain, treated with level 3 analgesic and / or already treated for neuropathic pain
* Drug-addicted patients
* Pregnant or lactating women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with major functional surgery associated with moderate-to severe postoperative pain in the enhanced recovery settings.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
System Usability Score | 72 hours after use of Zalviso
  A 10 items Licket type System Usability Score will be used in patients with ZALVISO® analgesia and in carrying ward nurses 72 hours the surgery per each case.

SECONDARY OUTCOMES:
Satisfaction Score | 72 hours after use of Zalviso
  100 points (0 - no satisfaction; 100 - entire satisfaction) satisfaction score will be used in physical therapist 72 hours after the surgery per each case.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric AUBRUN, MD, PhD, Principal Investigator — Service d'Anesthésie Réanimation - Hôpital de la Croix-Rousse - Lyon; Mikhail DZIADZKO, MD, Principal Investigator — Service d'Anesthésie Réanimation - Hôpital de la Croix-Rousse - Lyon
Locations (1):
- Hôpital de la Croix Rousse - Service d'Anesthésie-Réanimation, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amson H, Lasselin P, Naegels B, Pardey Bracho GF, Aubrun F, Dziadzko M. Usability evaluation of sufentanil sublingual tablet analgesia in patients following Enhanced Recovery After Surgery. J Comp Eff Res. 2021 Jun;10(9):743-750. doi: 10.2217/cer-2020-0239. Epub 2021 Apr 21. PMID 33880939